CLINICAL TRIAL: NCT05757102
Title: A Phase 3, 24-week, Randomized, Double-blind, Parallel-group Bayesian Dynamic Borrowing Study Comparing the Efficacy, Safety, Tolerability and Pharmacokinetics of FF/UMEC/VI With FF/VI in 12-17-year-old Participants With Inadequately Controlled Asthma on Stable Maintenance Therapy With ICS/LABA
Brief Title: A Study to Compare the Efficacy, Safety and Tolerability of FF/UMEC/VI With FF/VI in 12-17-year-olds With Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206867
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Fluticasone Furoate; GW685698; Umeclidinium; GSK573719; Vilanterol; GW642444; Trelegy; Relvar; Breo
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving FF/UMEC/VI (Experimental)
  Interventions: Drug: FF/UMEC/VI; Device: ELLIPTA
- Participants receiving FF/VI (Active Comparator)
  Interventions: Device: ELLIPTA; Drug: FF/VI

INTERVENTIONS:
Drug: FF/UMEC/VI — FF/UMEC/VI will be administered.
  Arms: Participants receiving FF/UMEC/VI
Device: ELLIPTA — FF/UMEC/VI and FF/VI will be administered via ELLIPTA inhaler
Drug: FF/VI — FF/VI will be administered.
  Arms: Participants receiving FF/VI

SUMMARY:
The primary purpose of this study is to evaluate the effects of Fluticasone Furoate (FF)/ Umeclidinium (UMEC)/ Vilanterol (VI) on lung function compared with FF/VI after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 12 to 17 years of age (inclusive), at the time of signing the informed consent/assent.
* Participants who have a diagnosis of asthma as defined by the National Institutes of Health [NIH, 2020] at least 1 year prior to Visit 0.
* Participants who have required daily Inhaled corticosteroids (ICS)/ Long-Acting Beta2-Agonist (LABA) treatment for at least 12 weeks prior to Visit 0 with no changes to maintenance asthma medications during the 6 weeks immediately prior to Visit 0 (including no changes to a stable total ICS dose of >250 to <=500 microgram (mcg)/day fluticasone propionate, or equivalent).
* In the 1 year prior to Visit 1: A documented healthcare contact for acute asthma symptoms; OR A documented temporary change in asthma therapy for acute asthma symptoms, according to a prespecified asthma action plan (or equivalent).
* Participants with inadequately controlled asthma (ACQ-6 score ≥1.5) at Visit 1, despite ICS/LABA maintenance therapy.
* A best pre-bronchodilator FEV1 >40% to <=90% of the predicted normal value and a ≥12% increase in FEV1 with albuterol/salbutamol at Visit 1. Predicted values will be based on the European Respiratory Society (ERS) Global Lung Function Initiative.

Exclusion Criteria:

* Chest X-ray documented pneumonia in the 6 weeks prior to Visit 1.
* Any asthma exacerbation requiring a change in maintenance asthma therapy and/or the use of systemic corticosteroids for at least 3 days in the 6 weeks prior to Visit 1. (Participants requiring a temporary change in asthma therapy (e.g., oral corticosteroids or increased dose of ICS) to treat an exacerbation in the 6 weeks prior to Visit 1 are not explicitly excluded at Visit 1 provided that, at the Investigator's discretion, the participant's condition is stable after they have resumed their pre-exacerbation maintenance asthma therapy (without modification), returned to their baseline asthma status and they are considered appropriate for enrollment into this study of up to 6 months duration)
* History of Life-threatening Asthma
* Participants with current evidence of active pulmonary diseases or abnormalities other than asthma (e.g., pneumonia, active tuberculosis, significant bronchiectasis, etc.).
* Current smokers and users of other inhaled products for recreation with or without nicotine (defined as participants who use cigarettes, e-cigarettes, other/vaping-related devices, cigars or pipe tobacco]) within 12 months prior to Visit 1.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 292 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in trough forced expiratory volume in 1 second (FEV1) (Liters) at Week 24 | Baseline (Week 0) and Week 24
  FEV1 will be measured using spirometry.

SECONDARY OUTCOMES:
Change from Baseline in Asthma Control Questionnaire (7 items) (ACQ-7) (Scores on a scale) | Baseline (Week 0) and Week 24
  ACQ-7 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation)), a question on rescue use and an additional item relating to lung function which is calculated based on FEV1. A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma.
Change from Baseline in Asthma Control Questionnaire (6 items) (ACQ-6) (Scores on a scale) | Baseline (Week 0) and Week 24
  ACQ-6 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation)) and a question on rescue bronchodilator use. A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma.
Change from Baseline in Asthma Control Questionnaire (5 items) (ACQ-5) (Scores on a scale) | Baseline (Week 0) and Week 24
  ACQ-5 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation). A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma.
Number of Participants with a clinically important change from baseline in ACQ-7 Score | Week 24
  ACQ-7 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation)), a question on rescue use and an additional item relating to lung function which is calculated based on FEV1. A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma. A change of 0.5 in score suggests a clinically important change in score.
Number of Participants with a clinically important change from baseline in ACQ-6 Score | Week 24
  ACQ-6 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation)) and a question on rescue bronchodilator use. A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma. A change of 0.5 in score suggests a clinically important change in score.
Number of Participants with a clinically important change from baseline in ACQ-5 Score | Week 24
  ACQ-5 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation). A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma. A change of 0.5 in score suggests a clinically important change in score.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (26):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Paradise Valley, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Waco, Texas
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (2):
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Joondalup WA, Western Australia
- GSK Investigational Site, Santiago, Chile
- GSK Investigational Site, Ebdentown, New Zealand
- South Korea (3):
  - GSK Investigational Site, Cheongju Chungcheongbuk-do
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/